CLINICAL TRIAL: NCT01686659
Title: Noninvasive and Continuous Hemoglobin Monitoring for Surgical Blood Management
Acronym: NACHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Society for the Advancement of Blood Management, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NACHO
Record Dates: First submitted 2012-08-29; First posted 2012-09-18 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Surgery
Keywords: Transfusion; Continuous Hemoglobin Monitoring; SpHb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SpHb Arm (Experimental): These are the patients whose primary anesthesiologists have been allocated to treat them while having access to data from a continuous noninvasive hemoglobin monitoring device
  Interventions: Device: Continuous Noninvasive Hemoglobin Monitoring
- Control Arm (No Intervention): These are the patients whose primary anesthesiologists have been allocated to treat them without having access to data from a continuous noninvasive hemoglobin monitoring device

INTERVENTIONS:
Device: Continuous Noninvasive Hemoglobin Monitoring — Availability of data from a continuous noninvasive hemoglobin monitoring device (total hemoglobin [SpHb] and Pleth Variability Index [PVI]) to the clinicians in the operating room
  Other Names: SpHb; Radical-7; Radical 7 Pulse CO-Oximeter
  Arms: SpHb Arm

SUMMARY:
This is a multi-center cluster-randomized trial with the following Specific Aims:

* To evaluate if continuous noninvasive hemoglobin monitoring will reduce the RBC transfusions in patients undergoing surgeries associated with a significant risk of bleeding.
* To evaluate if patients monitored with continuous noninvasive hemoglobin experience less frequent complications and shorter hospital stay compared with patients who are not being monitored with continuous noninvasive hemoglobin.

Accordingly, the study hypotheses are defined as follows:

* The primary null hypothesis is that continuous noninvasive hemoglobin monitoring will not reduce the RBC transfusions in patients undergoing surgeries associated with a significant risk of bleeding.
* The secondary hypothesis is that in patients monitored with continuous noninvasive hemoglobin, there will be earlier warning of critical drops in hemoglobin, and thus, there will be less frequent complications compared with patients who are not being monitored with continuous noninvasive hemoglobin.

DETAILED DESCRIPTION:
This is a matched-pair cluster-randomized controlled trial. At each participating centers, consenting eligible Anesthesiologists will be grouped into matched pairs based on their practice characteristics and experience (namely, their main surgical service/procedures and their years of experience working as a clinician responsible for making transfusion decisions). From each pair, Anesthesiologists will be randomly allocated to either treat their patients while having access to data from a continuous noninvasive hemoglobin monitoring device (total hemoglobin [SpHb] and Pleth Variability Index [PVI]) (SpHb group) or without access to SpHb/PVI data, under standard of care (control group). Regardless of randomization, all patients will be monitored with the device but the data will be blinded and not be available to the Anesthesiologist to be used in the management of the control group. Only in the SpHb group, the SpHb/PVI data will be provided live to the Anesthesiologist, to be used during management of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing one of the listed major surgeries associated with possibility of significant blood loss
* Consenting patients who are primarily managed by the consenting Anesthesiologists participating in the study (Not applicable at participating centers which have obtained a waiver of informed consent for the patients from their respective IRB)
* At least one finger available and accessible for performing non-invasive hemoglobin monitoring (preoperative perfusion index greater than 0.5)

Exclusion Criteria:

* Any patients who do not fit the criteria for use of sensor, specifically, any patient with nail polish and/or a nail deformity, or obstructed physical access (e.g. due to bandage) to all fingers that would be used for sensor placement, in a manner that interferes with satisfactory sensor placement
* Any patients being monitored with motor evoked potential devices
* Any patients with a known hemoglobinopathy
* Any patients undergoing Cardio-Pulmonary Bypass (CPB)
* Any patients who cannot be transfused or has refused consent for a blood transfusion
* Patients who are moribund/salvage cases as determined by the participating Anesthesiologist in charge of management of the patient in the operating room
* Patients being treated by any artificial oxygen carriers within 30 days of hospital stay
* Patients who are actively enrolled in or within 30 days of completion of any other study (except for purely observational studies with no intervention)
* Patients being managed outside of an operating room in the participating centers, or in operating room with conditions not conducive to perform and complete the study procedures (including use of the hemoglobin monitoring device)
* Patients younger than 18 years old
* Patients who are pregnant
* Any patients expected to receive transfusion preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Amount of Intraoperative RBC Transfusion | From the first surgical incision to the wound closure
  Number of allogeneic RBC units transfused intraoperatively per patient

SECONDARY OUTCOMES:
Intraoperative RBC Transfusion Rate | From the first surgical incision to the wound closure
  Occurrence of any allogeneic RBC transfusions intraoperatively
Amount of Perioperative RBC Transfusion | From time of admission to the hospital to the time of discharge or death whichever sooner (an estimated average of 6 days)
  Total number of allogeneic RBC units transfused perioperatively during hospital stay
Ischemic Events | From time of surgery to the time of discharge or death whichever sooner (an estimated average of 5 days)
  Incidence of new (or worsening of pre-existing) ischemic events
Mortality | From time of surgery to 30 days after the surgery
  Any death occuring during surgery or within 30-day period following the surgery
Length of Stay | From time of surgery to time of discharge from hospital (an estimated average of 5 days)
  Length of post-surgery hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Aryeh Shander, MD, Principal Investigator — Englewood Hospital & Medical Center; Mazyar Javidroozi, MD, PhD, Study Director — Englewood Hospital & Medical Center; Aryeh Shander, MD, Study Chair — Englewood Hospital & Medical Center
Locations (8):
- United States (5):
  - Stanford University, Stanford, California
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Swedish Medical Center, Seattle, Washington
- CHU Angers, Angers, France
- IRCCS Policlinico San Donato, San Donato, MI, Italy
- Sapporo Medical University School of Medicine, Chuo-ku Sapporo, Hokkaido, Japan